CLINICAL TRIAL: NCT06151730
Title: Hypertension Management and Cardiovascular Adverse Event Prevention in Patients With B-Cell Malignancies Undergoing Treatment With Bruton Tyrosine Kinase Inhibitors (HALT) - A Pilot Study
Brief Title: Evaluation of Hypertension Management and Cardiovascular Adverse Event Prevention in Patients With B-cell Malignancies Undergoing Treatment With Bruton Tyrosine Kinase Inhibitors, the HALT Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joerg Herrmann, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 23-007083; NCI-2023-09519 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-007083 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia; Hematopoietic and Lymphoid System Neoplasm; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients attend hypertension clinic visits, undergo optional blood pressure monitoring, electrocardiograms, impedance cardiography testing and blood and urine sample collection and have medical records reviewed throughout study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the incidence and management of new and worsening high blood pressure in patients with B-cell cancers on BTKi treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively define the incidence of new and/or worsening HTN in patients with B-cell malignancies on BTKi.

II. To identify the hemodynamic changes associated with new and/or worsening HTN in patients with B-cell malignancies on BTKi by impedance cardiography (ICG) and thereby to define the optimal anti-hypertensive strategies.

III. To compare 1-year MACE rates between patients with B cell malignancies on BTKi with new or worsening HTN on optimal anti-HTN strategies with patients who do not develop HTN on BTKis.

OUTLINE: This is an observational study.

Patients attend hypertension clinic visits, undergo optional blood pressure monitoring, electrocardiograms, impedance cardiography testing and blood and urine sample collection and have medical records reviewed throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lymphocytic leukemia (CLL), mantle cell lymphoma (MCL), Waldenstrom macroglobulinemia (WM), and marginal zone lymphoma (MZL), planned to begin Bruton tyrosine kinase inhibitors (BTKi) treatment or who will start a new BTKi agent after a 5-day wash out period (either as a single agent or on combination with other chemotherapies), who are willing to return to Mayo Clinic for ongoing follow-up

Exclusion Criteria:

* Patients with known central nervous system (CNS) involvement of their B-cell malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with B-cell malignancies on BTKi treatment at Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular events (MACE) | Up to 12 months
  1-year MACE rates between patients with B-cell malignancies on BTKi with new or worsening HTN on optimal anti-HTN strategies will be compared with patients who do not develop HTN on BTKi.

SECONDARY OUTCOMES:
Incidence of new and/or worsening hypertension (HTN) | Up to 12 months
  Incidence of new or worsening HTN over 1 year of BTKi therapy will be recorded (defined as blood pressure (BP) increase to>140 mmHg systolic or > 90 mmHg diastolic).
Hemodynamic changes associated with new and/or worsening HTN | Up to 12 months
  Impedance cardiography (ICG) changes from before to after BTKi initiation and anti-HTN therapy implication will be recorded to assess hemodynamic changes.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Herrmann, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials